CLINICAL TRIAL: NCT02205983
Title: The Effects of Hydromorphone on Responses to Verbal Tasks
Acronym: HESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: UC13-1027; R01DA002812 (NIH)
Record Dates: First submitted 2014-07-28; First posted 2014-08-01 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-09

CONDITIONS: Healthy
Keywords: enrolling; adult; volunteers
MeSH Terms: interventions — Hydromorphone; Acetaminophen; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 2 mg hydromophone (Experimental): Healthy adult volunteers will receive 2 mg hydromophone. Hydromorphone is a mu-opioid agonist used clinically for pain management. Plasma concentrations of hydromorphone peak approximately 60 min after ingestion.
  Interventions: Drug: 2 mg hydromorphone
- 4 mg hydromphone (Experimental): Healthy adult volunteers will receive 4 mg hydromophone. Hydromorphone is a mu-opioid agonist used clinically for pain management. Plasma concentrations of hydromorphone peak approximately 60 min after ingestion
  Interventions: Drug: 4 mg hydromorphone
- 1000 mg acetaminophen (Experimental): Healthy adult volunteers will receive 1000 mg acetaminophen. Acetaminophen is a COX inhibitor that is used clinically as an analgesic and antipyretic. The dose administered here has been shown to reduce neural and subjective responses to social rejection, and it also peaks about 60 min after ingestion.
  Interventions: Drug: 1000 mg Acetaminophen
- Dextrose (Placebo Comparator): Healthy adult volunteers will recieve Dextrose (placebo).
  Interventions: Drug: dextrose

INTERVENTIONS:
Drug: 2 mg hydromorphone — We are administering oral hydromorphone to healthy volunteers to measure its effects on the performance of a verbal task.
  Arms: 2 mg hydromophone
Drug: 1000 mg Acetaminophen — We are administering sublingual buprenorphine to healthy volunteers to measure its effects on the performance of a verbal task.
  Arms: 1000 mg acetaminophen
Drug: 4 mg hydromorphone — We are administering oral hydromorphone to healthy volunteers to measure its effects on the performance of a verbal task.
  Arms: 4 mg hydromphone
Drug: dextrose — We are administering dextrose to healthy volunteers for our placebo group.
  Arms: Dextrose

SUMMARY:
In this study, the investigators will examine the effects of hydromorphone, as compared to placebo, upon physiological, subjective, and hormonal responses to a stressful speech task and a non-stressful control task in healthy adults. There is strong evidence in support of the role of endogenous opioids and opiates in mediating social behavior in humans and other animals, and particularly, in social distress. The investigators have recently shown that buprenorphine, a partial mu-opioid agonist, reduces cortisol responses to stress. Here, the investigators propose to further explore the role of the opioid system in mediating stress responses in humans through the use of hydromorphone, a full mu opioid agonist, in addition to acetaminophen. The investigators hypothesize that like acetaminophen, hydromorphone will reduce both physiological and subjective measures of stress.

DETAILED DESCRIPTION:
Participants be randomly assigned to receive 1000 mg acetaminophen, 2mg hydromorphone, 4mg hydromorphone, or placebo at each of two sessions; one during which they well participate in a stressful speaking task, and one during which they'll participate in a nonstressful control task. Physiological and subjective measures will be taken throughout each session.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers

Exclusion Criteria:

1. any current medical condition requiring medication or abnormal electrocardiogram
2. current or past medical condition considered to be a contraindication for the study conditions
3. any current Axis I psychiatric disorder (APA, 1994) including Substance Use Disorder, or Anxiety Disorder or Major Depression in the past year, any history of psychosis
4. less than high school education
5. lack of fluency in English
6. night shift work
7. Pregnancy, lactation or plans to become pregnant.
8. Use of hormonal contraception.
9. Daily cigarette smokers i.e., >7 cigarettes per week

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harriet de Wit, PhD, Principal Investigator — University of Chicago; Jerome Jaffe, MD, Study Chair — University of Maryland
Locations (1):
- University of Chicago Hospital, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were excluded if they had a serious medical condition, abnormal electrocardiogram, Axis I psychiatric disorder in the past year, or a history of psychosis. Subjects were also excluded if they had not completed high school, were not fluent in English, worked a night shift, used hormonal contraceptives, or were pregnant.
Period: Overall Study
Arm/Group | 2 mg Hydromorphone | 4 mg Hydromorphone | 1000 mg Acetaminophen | Dextrose (Placebo)
Started | 12 | 12 | 13 | 13
Completed | 12 | 12 | 13 | 13
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 4 mg Hydromorphone: Healthy adult volunteers will receive 4 mg hydromophone. Hydromorphone is a mu-opioid agonist used clinically for pain management. Plasma concentrations of hydromorphone peak approximately 60 min after ingestion
- Dextrose (Placebo): Healthy adult volunteers will receive Dextrose (placebo).
- Total: Total of all reporting groups
Arm/Group | 2 mg Hydromophone | 4 mg Hydromorphone | 1000 mg Acetaminophen | Dextrose (Placebo) | Total
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Row population differs from overall as demographic characteristics of participants is broken down by which group they were randomized into.
  years | 19.9 (1.8) | 21.2 (2.8) | 23.6 (6.6) | 23.1 (4.4) | 22 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Row population differs from overall as demographic characteristics of participants is broken down by which group they were randomized into.
  Participants
    Female | 4 | 4 | 6 | 5 | 19
    Male | 8 | 8 | 7 | 8 | 31
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 13 | 13 | 50

OUTCOME MEASURES:

1. Primary Outcome: Subjective Effects as Assessed by Score on "Feel Drug", "Feel High", "Like Drug", and "Want More" Subscales of the Drug Effects Questionnaire
Description: The Drug Effects Questionnaire (DEQ) is a visual analog scale questionnaire that assesses the extent to which subjects experience four subjective states: "Feel Drug", "Feel High", "Like Drug", and "Want More". The "Feel Drug", "Feel High", "Like Drug", and "Want More" subscales are reported. All subscales are scored on a visual analogue scale (scroll bar on computer screen) ranging from 0-100. 100 represents the highest score for that subjective state, and the higher the score, the worse the outcome. The values shown below are only from week 4
Time Frame: End of study (time 0 and approximately 4 weeks later), week 4 reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 2 mg Hydromophone | 4 mg Hydromphone | 1000 mg Acetaminophen | Dextrose
Number analyzed (Participants) | 12 | 12 | 13 | 13
units on a scale
  Feel Drug | 7.41 (1.2) | 14.75 (1.9) | 28 (1.5) | 5.76 (1.1)
  Like Drug | 25.9 (1.8) | 35.58 (2.5) | 9.61 (2.2) | 4.15 (1.4)
  Feel High | 6.08 (1.5) | 10.33 (1.01) | 15 (1.8) | 2.61 (1.8)
  Want More | 8.0 (2.1) | 26.83 (1.5) | 7.38 (1.96) | 2.65 (1.5)

ADVERSE EVENTS:
Arm/Group | 2 mg Hydromophone | 4 mg Hydromphone | 1000 mg Acetaminophen | Dextrose
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes